CLINICAL TRIAL: NCT01808586
Title: Facet Versus Trigger Point Injection for Management of Chronic Muscular Neck Pain: A Randomized Clinical Trial and Creation of a Clinical Prediction Algorithm
Brief Title: Facet Versus Trigger Point Injections for Chronic Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Dave Walton, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2982
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Neck Pain
Keywords: Neck; chronic pain; facet injection
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Betamethasone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexamethasone (Experimental): Intra-articular corticosteroid number 2.
  Interventions: Procedure: Dexamethasone
- Betamethasone (Experimental): Subjects will receive either betamethasone or dexamethasone injected into the cervical facet joints (levels determined by experienced physician).
  Interventions: Procedure: Betamethasone
- Intramuscular injection (Active Comparator): Subjects in this group will receive lidocaine injection directly into tender myofascial trigger points.
  Interventions: Procedure: Intramuscular Lidocaine
- Home exercise (Active Comparator): Subjects in this group will receive education and a pamphlet on a set of standardized home exercises for neck pain
  Interventions: Behavioral: Home Exercise

INTERVENTIONS:
Procedure: Betamethasone — 6 mg/mL injected into the facet joint as dictated by modified dual-comparative medial branch block diagnostic protocol
  Other Names: Betaject/Celestone
  Arms: Betamethasone
Procedure: Dexamethasone — 4mg/mL
  Arms: Dexamethasone
Procedure: Intramuscular Lidocaine — 2%
  Arms: Intramuscular injection
Behavioral: Home Exercise — Standardized home exercise program
  Arms: Home exercise

SUMMARY:
A) Background Chronic neck pain is a significant and common issue which is difficult to treat. Tight bands of muscle (trigger points) can be a source of chronic neck pain and they are sometimes injected to manage chronic neck pain. However, these injections seldom lead to significant, long-lasting relief. In some cases, these trigger points may originate from injury or damage to a specific joint in the neck (the facet joint). Treatment of this joint with cortisone injection may lead to improved pain relief and function.

B) Hypothesis By injecting the facet joint with cortisone, the pain associated with tight bands of muscle in the neck and shoulders will be relieved to a greater extent than that attained through trigger point injection.

C) Methods Patients with neck pain will have a test to determine if any pain originates from the facet joint. Among those who have significant pain from these joints, a comparison between the effect of cortisone injection into these joints versus injection into the trigger points will be evaluated.

D) Expected Results and Significance

It is expected that injection with cortisone into the facet joints will lead to improved pain and function when compared to that attained from trigger point injection. In addition, the number of trigger points, and the pain and headache that originate from these trigger points, are expected to decrease with cortisone injection into the facets to a statistically and clinically significant extent. Results from this pilot study will then influence the design of future trials into chronic neck pain treatment, leading to better clinical recommendations. A peer-reviewed publication and conference presentations will facilitate dissemination.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age and able to speak and understand conversational English
* Primary diagnosis of chronic (>6 months) mechanical / myofascial neck pain

Exclusion Criteria:

* Those with significant cognitive decline or cognitive interference (as identified by the physician) will be excluded, as will those who have received radiofrequency ablation of any cervical nerve within the past year, intra-articular cortisone facet injection within the past 4 months, trigger point injection into the cervical/shoulder girdle muscles within the past 4 months, or the presence of any known contraindication to injection (Attachments).
* Women who are or may be pregnant (based on last menstruation) will be excluded.
* Finally, for the purposes of this pilot study, those currently involved in active litigation regarding the neck pain will be excluded. Those with active worker's compensation claims or currently receiving salary indemnity benefits through motor vehicle insurance providers will be included, as they represent a significant proportion of this population.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Change (PGIC) | 1, 3, and 6 months
  A 15-point self-report scale ranging from 0 = A very great deal worse to 15 = A very great deal better (8 = no change).

SECONDARY OUTCOMES:
Pain Intensity Numeric Rating Scale | 1, 3, and 6 months
Neck Disability Index | 1, 3, and 6 months
Headache Impact Test - 6 | 1, 3, and 6 months
Patient Health Questionnaire - 9 | 1, 3, and 6 months
Adverse Events Checklist | 1, 3, and 6 months
  Constructed specifically for this study.
Global Cervical Active Range of Motion | 1, 3, and 6 months
  Measured using a digital inclinometer
Mechanical (Pressure) Pain Threshold | 1, 3, and 6 months
  Measured using a digital algometer over standardized myofascial trigger points.

CONTACTS AND LOCATIONS:
Overall Officials: David M Walton, BScPT, PhD, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Hospital / Parkwood Hospital, London, Ontario, Canada